CLINICAL TRIAL: NCT05235451
Title: Human-Animal Interactions to Improve Reading for Children With or at Risk for Learning Differences
Brief Title: Human-Animal Interactions to Improve Reading for Children With Learning Differences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Terrah Akard, Associate Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB #212366
Record Dates: First submitted 2022-01-20; First posted 2022-02-11 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Animal-Human Bonding; Learning Problem; Child Development
Keywords: Children with learning differences; Animal-assisted intervention
MeSH Terms: conditions — Human-Animal Bond

STUDY DESIGN:
Intervention Model Description: Children among 4 reading groups will be randomly assigned to a HAI intervention or control group. The 2 HAI intervention reading groups will receive visits from a registered canine team during children's small group reading sessions twice a week over 12 weeks. The 2 control reading groups will receive care as usual and offered a 1-time visit from the dog at the end of the study (after T3 completed).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The 2 HAI intervention reading groups will receive visits from a registered canine team during children's small group reading sessions twice a week over 12 weeks.
  Interventions: Other: Human-Animal Interactions
- Control group (No Intervention): The 2 control reading groups will receive care as usual and offered a 1-time visit from the dog at the end of the study (after T3 completed).

INTERVENTIONS:
Other: Human-Animal Interactions — Human-animal interactions (HAI) is a powerful and cost-effective strategy to improve reading fluencies and comprehension of children with learning differences. Emerging data suggest that HAI help promote classroom behaviors and learning, including effects on cognition, emotional functioning, and motor skills for children with and without learning differences. The HAI reading group will receive reading instruction as usual plus visits from a registered therapy dog team (dog + animal handler) twice a week over 12 weeks.
  Arms: Intervention group

SUMMARY:
The overall purpose of this study is to determine feasibility and preliminary efficacy of pet therapy, or human-animal interactions (HAI), for children (5-12 years of age) with or at risk for LD. Children among 4 reading groups will be randomly assigned to a HAI intervention or control group. The 2 HAI intervention reading groups will receive visits from a registered canine team during children's small group reading sessions twice a week over 12 weeks. The 2 control reading groups will receive care as usual and offered a 1-time visit from the dog at the end of the study (after T3 completed). Two weeks of initial work will focus on preliminary modifications to the protocol. Parents will complete electronic measures of psychological outcomes (child depression, anxiety, QOL) via REDCap at baseline (T1), 2 weeks post-baseline (T2), and 12 weeks post-baseline (T3). The investigators will obtain copies of reading assessments already conducted by the teachers at T1 and T3. Children's salivary cortisol will be obtained from participants in the intervention groups at T1, T2, and T3. Children and their parents will complete concluding interviews at study end (T3) to further inform what they liked and did not like about the intervention. Results of the proposed study will provide critical data for a future full-scale randomized clinical trial (R01) to examine the impact of HAI on psychological, physiological, and reading outcomes in children with or at risk for LD.

DETAILED DESCRIPTION:
According to the National Center for Learning Disabilities (NCLD), approximately 2.3 million children in the United States have learning differences (LD) such as dyslexia or ADHD. Despite improvement in educational interventions such as resource-room services and instructional styles, the availability of services to help these children and their families cope, adapt, and maintain quality of life (QOL) is inadequate. In particular, children with LD are especially at high risk for negative consequences, including both physical and mental health issues compared with typically developing children. Human-animal interactions (HAI) may be a powerful and cost-effective strategy to improve reading fluencies and comprehension of children with LD. Emerging data suggest that HAI help promote classroom behaviors and learning, including effects on cognition, emotional functioning, and motor skills for children with and without LD. Yet, empirical evidence using a rigorous approach to support the effectiveness of HAI with children with or at risk for LD is lacking. Previous studies endorse the effectiveness of HAI in promoting reading abilities and show promise to improve psychosocial outcomes for children, but have focused on typically developing children. No published studies have specifically targeted effects of HAI on children with or at risk for learning differences. More data are needed to substantiate positive effects on reading abilities associated with HAI. The long-term goal of this study is to improve reading abilities and reduce the negative psychological and social sequelae of children with learning differences (LD).

ELIGIBILITY:
<Inclusion Criteria>

Eligible Children are:

* 5-12 years of age
* With or at risk for a learning difference based on teacher report
* Assigned to a small reading group (approximately 3-5 children) that meets at least twice a week
* Able to understand English to complete consents and surveys
* Children both with and without dogs at home are allowed to participate in this study. Parents of subjects will be asked if they have a dog at home and, if so, to describe the child-dog relationship prior to data collection. This factor will be considered throughout the study
* Children taking medications are also allowed to participate in this study, and the investigators will consider medication protocols of subjects when evaluating outcomes.

Eligible Caregivers are:

* Parent or guardian as determined by person with whom each child resides for >50% of the time
* 18 years of age and up
* Able to understand English to complete consents and surveys

<Exclusion Criteria>

-Children self-reported fear of or allergies to canines.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-07-21 (Actual)

PRIMARY OUTCOMES:
Change in "Patient-Reported Outcomes Measurement Information System (PROMIS) Parent Proxy Scale v1.0 - Global Health 7" | Day 0, Day 84
  Child's overall quality of life before and after the intervention will be measured. This 5-point Likert scale measure (5=Excellent, 1=Poor) includes seven items. The final score could range from 7 to 35 and the higher scores mean higher quality of life.
Change in "Patient-Reported Outcomes Measurement Information System (PROMIS) Parent Proxy Short Form v1.1 - Depressive Symptoms 6b" | Day 0, Day 84
  Child's depressive symptoms before and after the intervention will be measured. This 5-point Likert scale measure (5=Almost Always, 1=Never) includes six items. The final score could range from 6 to 30 and the higher scores mean higher depressive symptoms.
Change in "Patient-Reported Outcomes Measurement Information System (PROMIS) Parent Proxy Short Form v2.0 - Anxiety 8a" | Day 0, Day 84
  Child's anxiety level before and after the intervention will be measured. This 5-point Likert scale measure (5=Almost Always, 1=Never) includes eight items. The final score could range from 8 to 40 and the higher scores mean higher anxiety level.
Change in "Child reading fluency" | Day 0, Day 84
  Copies of teacher evaluations of curriculum-based measure-oral reading fluency (e.g., CBM-ORF) already in use with the students will be obtained to measure reading fluency and comprehension at baseline (T1) and at the end of 12 weeks (T3) in both the intervention and control groups.
Change in "Child acute stress" | Day 0, Day 14, Day 84
  The investigators will measure salivary cortisol of child participants. Trained study staff will obtain salivary swabs from participants in the intervention groups before HAI begins (T1), after 2 weeks (T2), and at the conclusion of the study (T3). Saliva will be obtained and analyzed in the Vanderbilt Hormone Analytical Services Core.

SECONDARY OUTCOMES:
Satisfaction assessment after the intervention | Day 84
  End-of-study interviews will be conducted with children and parents in the intervention group to assess their satisfaction with the HAI.

CONTACTS AND LOCATIONS:
Overall Officials: Terrah F Akard, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Currey Ingram Academy, Brentwood, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
There are no tangible resources to share at this time as the intervention is in testing phases. The investigators plan to make the intervention available for sharing in the future, upon completed testing. Therefore, data is the only resource available for sharing.
  The proposed research will produce data with 40 children with or at risk for learning differences. The final data set will contain demographic information and children's psychological distress, acute stress, and reading fluency after the human-animal interaction.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available for sharing no later than the publication date of the main results from the final dataset. Data will be disclosed without a specific deadline.
Access Criteria: The data will be shared with anyone who is interested in this study. The investigators especially seek to make the data available to the community of scientists interested in human-animal interactions and their impact on children.